CLINICAL TRIAL: NCT03468751
Title: A Prospective Open-label Dose Escalation Phase 1 Study to Investigate the Safety and Tolerability, and to Determine the Maximum Tolerated Dose and Recommended Phase 2 Dose, of HLX10 in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study of HLX10, a Monoclonal Antibody Targeting Programmed Death-1 (PD-1) in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henlix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-001
Record Dates: First submitted 2018-03-11; First posted 2018-03-19 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor
Keywords: Metastatic; Refractory; Cancer; Solid; Tumor
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HLX10, Dose Finding Cohort (Experimental): Each cycle of treatment consists of 4 weeks. Patients who enroll into this study will receive an infusion of assigned dose of HLX10 once every two weeks. No intra-patient dose escalation is allowed. The proposed dose escalation sequence is 0.3, 1.0, 3.0, and 10 mg/kg, starting from 0.3 mg/kg.
  Interventions: Drug: HLX10
- HLX10, Dose Expansion Cohort (200 mg ) (Experimental): Each cycle of treatment consists of 4 weeks. Patients who enroll into this expansion cohort will receive an infusion of assigned dose of HLX10 at 200 mg once every two weeks.
  Interventions: Drug: HLX10

INTERVENTIONS:
Drug: HLX10 — recombinant humanized anti-PD-1 monoclonal antibody against solid cancers
  Other Names: anti-PD-1 monoclonal antibody

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of humanized anti-PD-1 monoclonal antibody, HLX10, in patients with advanced or metastatic tumors refractory to standard therapy. This study will also evaluate the pharmacokinetics, pharmacodynamics, immunogenicity and anti-tumor effect of HLX10 and explore the potential prognostic and predictive biomarkers.

DETAILED DESCRIPTION:
The lack of immunologic control is currently recognized as one of the hallmarks of cancer. The cancer immunoediting concept has been proposed as a mechanism by which tumors escape control. The concept involves three phases: elimination (tumor cell eradication), equilibrium (when editing of surviving tumor cells occurs) and escape (when the altered tumor cells progress through the shield of the activated immune response).

When the TCR of a T cell recognizes antigens expressed in the context of the MHC, the immune checkpoint modulates signaling: co-stimulatory molecules such as CD28 on T cells enhance the signal, whereas co-inhibitory molecules suppress it. Recent research has implicated the expression of immunoinhibitory checkpoints such as CTL antigen 4 (CTLA-4) and programmed death protein 1 (PD-1) as potential mediators of the equilibrium and escape phases of cancer immunoediting described above. These molecules are expressed on activated T cells, but when they bind to ligands either on antigen-presenting cells (CTLA-4 binding to CD80/CD86) or tumor cells (PD-1 binding to PD-L1), they tend to shut down the anti-tumor response. Efforts to use antibodies to target and block these immuno-inhibitory interactions have ushered in a new era of immunotherapy.

Tumors display a wide variety of antigens that can potentially be exploited by harnessing the adaptive immune response. The T-cell response to these antigens can be dysregulated by tumor cells seeking to evade immunologic detection and destruction by hijacking physiological homeostatic immune-checkpoint signaling pathways. In addition to a variety of mechanisms that can create an immunosuppressive microenvironment (e.g. secretion of inhibitory cytokines, presence of regulatory T cells), many tumor types also express PD-L1.

Nivolumab and pembrolizumab are the two anti-PD1 monoclonal antibodies currently approved for multiple cancers. The application of nivolumab or pembrolizumab alone or in combination with chemotherapy has completely changed cancer management.

HLX10 is a new monoclonal antibody targeting PD1 on T cells, developed from mouse hybridoma technology. In vitro studies have demonstrated the growth inhibition of multiple cancer cell lines, and shown growth inhibition of tumors in murine xenogeneic studies.

Nonclinical studies dosing up to 50 mg/kg HLX10 weekly in cynomolgus monkeys for 13 weeks have shown good tolerability without evident toxicities (please refer to Investigator's Brochure). HLX10 shows cross-reactivity to both monkey and human PD1, but does not bind rodent PD1.

Based on the pharmacology studies and pharmacokinetic and toxicokinetic studies in cynomolgus monkeys, this study is a phase-1 study to address the safety and tolerability of HLX10 in patients with metastatic or recurrent cancer.

HLX10 has not yet been tested in human. Therefore, the investigators propose this first-in-human phase 1 study. In this study, the investigators intend to investigate the safety, and tolerability of HLX10 in humans, and hope to identify the maximum tolerated dose (MTD), and determine the recommended phase 2 dose in future study. At the same time, the investigators would like to gain information of the pharmacokinetics and pharmacodynamics of this drug and its potential immunogenicity.

To minimize the risk of patients who volunteer to receive this experimental drug, the investigators will choose 0.1 mg/kg as the initial starting dose. The selection of starting dose is based on the repeat-dose toxicology study on monkey, at 1/166 of the human equivalent dose of No-Observed Adverse Effect Level (NOAEL) in cynomolgus studies.

To investigate the dose required to reach maximal effect, the investigators propose a dose escalation sequence. The purpose of the dose escalation is to obtain the pharmacokinetics and pharmacodynamics of HLX10 at different dose levels, and investigate its relationship with adverse reactions. The investigators also intend to identify the MTD. The information from the dose escalation is crucial to determine the optimal dose in future studies and potential indications for HLX10.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed, unidimensionally-measurable and/or evaluable carcinoma which has failed standard therapy or for which no standard therapy is available.
2. ECOG performance status score of ≤ 2 at study entry.
3. Able to provide written informed consent.
4. A life expectancy longer than three months as determined by the investigator.
5. Adequate hematologic functions, as defined by: absolute neutrophil counts ≥ 1500/mm3; a hemoglobin level ≥ 10 gm/dL; a platelet count ≥ 100,000/mm3.
6. Adequate hepatic function defined by: a total bilirubin level ≤ 1.5x of upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x of ULN or ≤ 5x of ULN in known hepatic metastases or with primary hepatocellular carcinoma.
7. Adequate renal function, as defined by the creatinine clearance rate ≥ 50 mL/minute by Cockcroft-Gault formula.
8. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥ 50%.
9. Use of effective contraceptive measures if procreative potential exists.
10. At least 28 days from prior major surgery, prior cytotoxic chemotherapy, or prior therapy with investigational agents (or medical device) or local radiotherapy and at least 42 days from the last infusion of immune check point inhibitors (including anti-PD-1 or anti-PD-L1) before the first infusion of investigational product.
11. For patients with hepatocellular carcinoma, their Child-Pugh score has to be A.
12. Able to be followed up as required by the study protocol.

Exclusion Criteria:

1. Patients who still have persistent ≥ grade 2 toxicities from prior therapies.
2. Concurrent unstable or uncontrolled medical conditions. Either of the followings:

   * Active systemic infections;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥100 mmHg), or poor compliance with anti-hypertensive agents;
   * Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (class III or IV of New York Heart Association [NYHA]) or acute myocardial infarction within 6 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemic agents;
   * The presence of chronically unhealed wound or ulcers;
   * Other chronic diseases, which, in the opinion of the investigator, could compromise safety of the patient or the integrity of study.
3. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not taking steroids for brain edema). Anticonvulsants are allowed.
4. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 3 years are allowed to participate).
5. Pregnancy (confirmed by serum beta human chorionic gonadotropin [ßHCG]) or breast-feeding.
6. Known history of human immunodeficiency virus infection (HIV).
7. Patient who has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroid (more than 10 mg per day) or immunosuppressive agents.
8. Patient who has active hepatitis B (HBsAg reactive) or hepatitis C (defined anti-HCV reactive)
9. Patient who has a history of interstitial lung disease
10. The patient is the investigator, sub-investigator or any one directly involved in the conduct of the study.
11. Patient has a history or current evidence of any condition or disease that could confound the results of the study, or is not the best interest of the patient to participate, in the opinion of Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Numbers and percentage of patients with adverse events (AEs) | 1 year
Maximum tolerated dose of HLX10 | 1 year

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of HLX10 in different cohorts. | 1 year
Minimum concentration (Cmin) of HLX10 in different cohorts. | 1 year
Area under concentration (AUC0-tau) in different cohorts. | 1 year
Half-life (T1/2) of HLX10 in different cohorts. | 1 year
Clearance (CL) rate of HLX10 in different cohorts. | 1 year
Volume of distribution (Vss) at steady state in different cohorts. | 1 year
The presence and percentage of anti-HLX10 antibody (immunogenicity). | 1 year
Disease control rate. | 1 year
Overall response rate. | 1 year
Duration of response. | 1 year
Receptor occupancy of PD-1 on human T cells. | 1 year
Potential predictive and prognostic biomarkers. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gi-Ming Lai, MD, Principal Investigator — Taipei Municipal Wanfang Hospital
Locations (1):
- Taipei Municipal Wanfang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho CL, Chao TY, Chang CL, Lin HY. Safety, Tolerability, and Preliminary Efficacy of Serplulimab, a Novel Anti-PD-1 Antibody, in Patients with Metastatic or Recurrent Solid Tumors: A Phase I Study. BioDrugs. 2024 Mar;38(2):287-299. doi: 10.1007/s40259-023-00639-w. Epub 2024 Jan 9. PMID 38194016